CLINICAL TRIAL: NCT06613399
Title: A Randomized Controlled Study of Multi-technology Integration Total Mesorectal Excision (MTI-TME) Versus Conventional Total Mesorectal Excision (C-TME) for the Treatment of Middle and Distal Rectal Cancer.
Brief Title: Multi-Technology Integrated Total Mesorectal Excision Versus Conventional Total Mesorectal Excision for the Treatment of Middle and Distal Rectal Cancer.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRSYM202409
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer
Keywords: MTI-TME; anastomotic leakage
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Technology Integrated Total Mesorectal Excision，MTI-TME (Experimental)
  Interventions: Procedure: MTI-TME
- Conventional Total Mesorectal Excision，C-TME (Placebo Comparator)
  Interventions: Procedure: C-TME

INTERVENTIONS:
Procedure: MTI-TME — Multi-Technology Tntegrated Total Mesorectal Excision，MTI-TME
  Arms: Multi-Technology Integrated Total Mesorectal Excision，MTI-TME
Procedure: C-TME — Conventional Total Mesorectal Excision，C-TME
  Arms: Conventional Total Mesorectal Excision，C-TME

SUMMARY:
A multicenter, prospective, randomized, controlled clinical trial of multi-technology integration total mesorectal excision (MTI-TME) versus conventional total mesorectal excision (C-TME) for the treatment of middle and distal rectal cancer

DETAILED DESCRIPTION:
Currently, laparoscopic total mesorectal excision (TME) has become the standard procedure for treating middle and distal rectal cancer. Anastomotic leakage has always been one of the serious complications of TME surgery, and Anastomotic leakage not only increases the hospital expenses, but also brings physical discomfort and psychological pain to the patients. Furthermore, anastomotic leakage is associated with a heightened risk of anastomotic stenosis, compromised bowel function, delayed initiation of postoperative adjuvant therapy, increased local recurrence rates post-surgery, and diminished long-term survival outcomes. A report from the Netherlands indicates that anastomotic leakage serves as an independent prognostic factor for overall survival in patients diagnosed with rectal cancer. Prior studies have documented the incidence of anastomotic leakage to range between 3.6% and 21%, attributable to a confluence of various factors including technical complications, oncological considerations, and the patient's overall health status. Among these determinants, aspects such as blood supply adequacy, tension at the site of anastomosis, tissue quality, and anatomical positioning of the rectum are widely recognized as significant risk factors for developing anastomotic leaks.Currently, several strategies are employed to mitigate the incidence of anastomotic leakage, including preoperative proctocolectomy, anal decompression placement, vertical transverse resection of the rectum, and anastomotic reinforcement techniques. In our clinical practice, we have innovatively integrated multiple approaches: (1) preservation of the left colic artery (LCA); (2) high-level resection of the inferior mesenteric vein (IMV); (3) standardized mobilization of the splenic flexure along with left lateral colon; (4) multi-plane dissection of mesorectal flaps; and (5) selective reinforcement at the anastomosis. Our findings indicate that multi-technology integrated total mesorectal excision (MTI-TME) significantly reduces both preventive stoma rates and incidences of anastomotic leakage compared to conventional total mesorectal excision (C-TME), . However, there remains a lack of robust evidence-based medicine supporting MTI-TME's advantages in treating middle and distal rectal cancer; further research is urgently needed to provide additional clinical evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged 18 to 75.
2. Histopathological examination of the preoperative biopsy confirms adenocarcinoma.
3. Preoperative MRI shows the tumor's lower margin is below the umbilical ligament.
4. High-resolution CT and MRI do not indicate suspicious distant metastasis.
5. Participants' general condition is acceptable, with an ASA score of ≤3 before surgery.
6. Participants must sign an informed consent form.

Exclusion Criteria:

1. Developing other malignant tumors within 5 years;
2. Multiple primary colorectal tumors;
3. Pregnant or lactating women;
4. Patients with severe mental disorders;
5. Severe intestinal diseases;
6. Poor general condition and uncontrolled comorbidities;
7. Ineligible for laparoscopic surgery;
8. Participating in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
anastomotic leakage rate | 1 year

SECONDARY OUTCOMES:
Operation time | During surgery
intraoperative blood loss | During surgery
3-year overall suvival rate | 3 years
local recurrance rate | 3 years
3-year disease-free survival rate | 3 years
3-year mortality rate | 3 years
postoperative quality of life | 3 years
  Postoperative quality of life will be evaluated by EORTC QLQ C30 Questionnaire
intestinal exhaust time | 1 year
postoperative pain | 1 year
  Postoperative pain will be assessed by numerical rating scale (NES).
colostomy rate | 1 year
hospital stay | 1 year
hospital cost | 1 year

IPD SHARING:
Plan to Share IPD: Undecided